CLINICAL TRIAL: NCT01168713
Title: A Randomized, Double-Blind, Multi-Center Study to Evaluate the Efficacy and Safety of Oral CEM-101 Compared to Oral Levofloxacin in the Treatment of Patients With Community-Acquired Bacterial Pneumonia
Brief Title: Efficacy and Safety Study of Oral CEM-101 Compared to Oral Levofloxacin in Treatment of Patients With Community-Acquired Bacterial Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE01-200
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Community-Acquired Bacterial Pneumonia
Keywords: Adults with Community-Acquired Bacterial Pneumonia
MeSH Terms: interventions — Levofloxacin; solithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levofloxacin (Active Comparator)
  Interventions: Drug: Levofloxacin
- CEM-101 (Experimental)
  Interventions: Drug: CEM-101

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin once daily for 5 days:
  Levofloxacin 750 mg PO Days 1-5
  Other Names: Levaquin
  Arms: Levofloxacin
Drug: CEM-101 — CEM-101 once daily for 5 days:
  CEM-101 800 mg PO Day 1
  CEM-101 400 mg PO Days 2-5
  Other Names: Solithromycin
  Arms: CEM-101

SUMMARY:
Study to evaluate the safety and efficacy of oral CEM-101 compared to oral Levofloxacin in the treatment of adults with moderate to moderately severe community-acquired bacterial pneumonia.

DETAILED DESCRIPTION:
Community-acquired bacterial pneumonia is an acute infection of the pulmonary parenchyma with symptoms such as fever or hypothermia, chills, rigors, chest pain, and/or dyspnea. The widespread emergence of antibiotic resistant pathogens, including the macrolide-resistant Streptococcus pneumoniae, has resulted in a need for new and effective antibiotics that have activity again CABP pathogens. CEM-101 is the first fluoroketolide with excellent in vitro and in vivo activity against resistant S. pneumoniae and other key typical and atypical bacterial respiratory pathogens.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of community acquired bacterial pneumonia (e.g. cough with purulent sputum or change in character of sputum consistent with bacterial infection, dyspnea or tachypnea, chest pain due to pneumonia, fever, presence of rales and/or signs of consolidation).
2. No prior systemic antibacterial therapy, unless failed other therapy.
3. Chest Xray shows new lobar or multilobar infiltrate(s) consistent with acute bacterial pneumonia.
4. PORT Risk Class II, III, or IV <=105
5. Ability to take oral medication.

Exclusion Criteria:

1. Severe chronic obstructive pulmonary disease FEV1 <30%.
2. Hospitalization within 90 days or residence in a long-term-care facility within 30 days prior to the onset of symptoms
3. Chemotherapy or radiation therapy within the previous 3 months.
4. Significant hepatic, hematological, renal abnormalities.
5. Any concomitant condition that, in the opinion of the Investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy and follow-up could be completed (e.g. life expectancy <30 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Clinical Success in the Intent to Treat (ITT) population at the Treatment of Cure (TOC) visit | 5 to 10 days after the last dose of study drug
  Clinical Success defined as continued improvement or complete resolution of baseline signs and symptoms and if available, an improved/stable chest radiograph after the end of treatment
Clinical Success in the Clinically Evaluable (CE) population at the Treatment of Cure (TOC) Visit | 5 to 10 days after the last dose of study drug
  Clinical Success defined as continued improvement or complete resolution of baseline signs and symptoms and if available, an improved/stable chest radiograph after the end of treatment

SECONDARY OUTCOMES:
By Patient Microbiological Response in the Microbiological Intent to Treat (microlITT) population at the end of treatment (EOT) | 5 days of study drug treatment
  Successful response is eradication, presumed eradication or combined eradication/presumed eradication of baseline pathogen.
By Patient Microbiological Response in the Microbiological Intent to Treat (microlITT) population at the Treatment of Cure (TOC) visit | 5 to 10 days after the last dose of study drug
  Successful response is eradication, presumed eradication or combined eradication/presumed eradication of baseline pathogen
By-patient Microbiological Response in the Microbiologically Evaluable (ME) populations at the end of treatment (EOT) | 5 days of study drug treatment
  Successful response is eradication, presumed eradication or combined eradication/presumed eradication of baseline pathogen
By-patient Microbiological Response in the Microbiologically Evaluable (ME) populations at Treatment of Cure (TOC) visit | 5 to 10 days after the last dose of study drug
  Successful response is eradication, presumed eradication or combined eradication/presumed eradication of baseline pathogen
Clinical Response in the Intent to Treat (ITT) population at End of Treatment (EOT) | 5 days of study drug treatment
  Clinical Success is defined as complete or near-complete resolution of the baseline signs and symptoms of community acquired bacterial pneumonia (CABP); no further study drug for treatment of CABP
Clinical Response in the microbiological intent to treat (microlITT) population at the end of treatment (EOT) | 5 days of study drug treatment
  Clinical Success is defined as complete or near-complete resolution of the baseline signs and symptoms of community acquired bacterial pneumonia (CABP); no further study drug for treatment of CABP
Clinical Response in the clinically evaluable (CE) population at the end of treatment (EOT) | 5 days of study drug treatment
  Clinical Success is defined as complete or near-complete resolution of the baseline signs and symptoms of community acquired bacterial pneumonia (CABP); no further study drug for treatment of CABP
Clinical REsponse in the Microbiologically Evaluable (ME) population at the end of treatment (EOT) | 5 days of study drug treatment
  Clinical Success is defined as complete or near-complete resolution of the baseline signs and symptoms of community acquired bacterial pneumonia (CABP); no further study drug for treatment of CABP
Early Clinical Response in the intent to treat (ITT) population at Day 3 | 3 days of study drug treatment
  Clinical success is defined as being both clinically stable and showing clinical improvement based on the symptoms of community acquired bacterial pneumonia (CABP)
Percentage of patients at each visit who have resolution of all baseline signs and symptoms in the clinically evaluable (CE) population | Day 3, Day 5 (end of treatment), and 5 to 10 days after the last dose of study drug (test of cure visit)
  Resolution of all baseline signs and symptoms in the clinically evaluable (CE) population
Percentage of patients at Day 3 who have resolution of cough, dyspnea, chest pain due to pneumonia and sputum production | 3 days of study drug treatment
  Resolution of cough, dyspnea, chest pain due to pneumonia and sputum production
Percentage of patients at the end of treatment (EOT) who have resolution of cough, dyspnea, chest pain due to pneumonia and sputum production | 5 days of study drug treatment
  resolution of cough, dyspnea, chest pain due to pneumonia and sputum production
Percentage of patients at Day 3 who are clinically stable | 3 days of study drug treatment
  clinical stability defined as:
  * Temperature <=37.8°C
  * Heart rate <=100 beats/min
  * Systolic blood pressure ≥90 mm Hg
  * Ability to maintain oral intake
  * Normal mental status (oriented to person, place or time)
Percentage of patients at the end of treatment (EOT) who are clinically stable | 5 days of study drug treatment
  Clinically stable defined as:
  * Temperature ≤37.8°C
  * Heart rate ≤100 beats/min
  * Systolic blood pressure ≥90 mm Hg
  * Ability to maintain oral intake
  * Normal mental status (oriented to person, place or time)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (44):
  - Birmingham, Alabama
  - Flagstaff, Arizona
  - Bell Gardens, California
  - Chula Vista, California
  - LeMesa, California
  - Los Angeles, California
  - Montclaire, California
  - Norwalk, California
  - Oceanside, California
  - Oxnard, California
  - Pasadena, California
  - Torrence, California
  - Waterbury, Connecticut
  - DeBary, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Kissimmee, Florida
  - Orlando, Florida
  - Blue Ridge, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Idaho Falls, Idaho
  - Morton, Illinois
  - Dubuque, Iowa
  - New Orleans, Louisiana
  - Fall River, Massachusetts
  - New Bedford, Massachusetts
  - Detroit, Michigan
  - Traverse City, Michigan
  - Butte, Montana
  - Las Vegas, Nevada
  - Akron, Ohio
  - Carlisle, Ohio
  - Eugene, Oregon
  - West Reading, Pennsylvania
  - Simpsonville, South Carolina
  - Rapid City, South Dakota
  - Franklin, Tennessee
  - Corsicana, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Draper, Utah
  - Magna, Utah
  - Salt Lake City, Utah
- Canada (8):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Saint-Jérôme, Quebec
  - Sherbrooke, Quebec
  - Trios-Rivieres, Quebec

REFERENCES:
- [Derived] Oldach D, Clark K, Schranz J, Das A, Craft JC, Scott D, Jamieson BD, Fernandes P. Randomized, double-blind, multicenter phase 2 study comparing the efficacy and safety of oral solithromycin (CEM-101) to those of oral levofloxacin in the treatment of patients with community-acquired bacterial pneumonia. Antimicrob Agents Chemother. 2013 Jun;57(6):2526-34. doi: 10.1128/AAC.00197-13. Epub 2013 Mar 18. PMID 23507282